# A See and Treat Paradigm for Cervical Pre-cancer

NCT02477124

Document Date: May 19, 2021

## **DUHS IRB Application (Version 1.10)**

| General Information |
|---|
| *Please enter the full title of your protocol: |
| A see and treat paradigm for cervical pre-cancer |
| *Please enter the Short Title you would like to use to reference the study: |
| A see and treat paradigm for cervical pre-cancer * This field allows you to enter an abbreviated version of the Study Title to quickly identify this study. |
| Add Study Organization(s): |
| List Study Organizations associated with this protocol: |
| Primary Department Name Department Name Dutts - Duke Default Department |
| Assign key study personnel (KSP) access to the protocol |
| * Please add a Principal Investigator for the study: (Note: Before this study application can be submitted, the PI MUST have completed CITI training) |
| Ramanujam, Nirmala |
| 3.1 If applicable, please select the Key Study personnel: (Note: Before this study application can be submitted, all Key Personnel MUST have completed CITI training) * Denotes roles that are not recognized in OnCore. Please select an appropriate role that is recognized in all clinical research applications (iRIS, OnCore, eREG, etc.) |
| A) Additional Investigators, Primary Study Coordinator (CRC), and the Primary Regulatory Coordinator (PRC): |
| Krieger, Marlee<br>Primary Regulatory Coordinator |
| B) All Other Key Personnel |
| Crouch, Brian Regulatory Coordinator Gallagher, Jennifer Study Coordinator (CRC/CRNC/RPL) Gonzales, Alana |

| Graduate Student Muasher, Lisa Collaborator Mueller, Jenna Research/Physician Assistant Skerrett, Erica Graduate Student Thiele, Bonnie Other | |
|---|---|
| *Please add a Study Contact: | |
| Krieger, Marlee Krieger, Marlee Ramanujam, Nirmala The Study Contact(s) will receive all important system notifications along with the Principal Investigator. (e.g., The study contact(s) are typically the Principal Investigator, Study Coordinator, and Regulatory Coordinator.) | |
| Oncore | |
| Please select the Library for your Protocol: | |
| This field is used in OnCore. Determines the Reference Lists, Forms, Protocol Annotations, Notifications, as Signoffs available for the protocol. Protocols that require reporting to the NCI (National Cancer Institute), select the Oncology library. Oncology Non-Oncology | |
| Protocol Application Type | |
| Select the type of protocol you are creating: | |
| <ul> <li>Please see additional criteria and information in the policy titled "Reliance on the IRB of Another Institution Organization, or an Independent IRB" on the IRB web site.</li> <li>Regular Study Application - Most common. The IRB will determine if the study is eligible for expeding review or requires full board review upon submission.</li> <li>Application for Exemption from IRB Review - Includes Exempt, Not Human Subject Research, &amp; Not Research.</li> <li>External IRB Application - Any study using an external IRB as the IRB-of-Record.</li> <li>Trainee Research While Away from Duke - Research conducted by medical students overseen by the Office of Curriculum &amp; other student/trainee research away from Duke.</li> <li>Individual Patient Expanded Access, Including Emergency Use - Use of an investigational product under expanded access, including emergency use of an investigational drug or biologic or emergency use of an unapproved device.</li> </ul> | lited<br>ot<br>the |
| Conflict of Interest | |
| Do any of the participating study investigators or other key personnel (or their immediate far other) have a financial or intellectual interest in, or are receiving compensation from, the spodrugs, devices or technologies used in this research? | |
| ⊙ Yes ○ No | |

| Has this conflict been disclosed to the Duke COI Committee? | |
|---|---|
| ⊙ Yes ○ No | |
| Are any key personnel an inventor of any of the drugs, devices or technologies used in this research? | |
| Have you filed an Inventor Disclosure Form? | |
| ⊙ Yes O No | |
| Do any key personnel have or anticipate (within the year) any financial relationships (e.g., consulting, speaking, advisory boards, patents, equity, options) that could be perceived to overlap or present a coof interest with the current research? | |
| O Yes ⊙ No | |
| Do any key personnel have a conflict of interest management plan or cautionary memo issued by DOS related to this research? | I-COI |
| ⊙ Yes ○ No | |
| If Yes, please give the name(s) of the relevant personnel. | |
| Nimmi Ramanujam | |
| Oversight Organization Selection | |
| Oversight Organization Selection CRU (Clinical Research Unit) or Oversight Organization Selection: | |
| CRU (Clinical Research Unit) or Oversight Organization Selection: | |
| CRU (Clinical Research Unit) or Oversight Organization Selection: Please select the CRU. OB/GYN | |
| CRU (Clinical Research Unit) or Oversight Organization Selection: Please select the CRU. | |
| CRU (Clinical Research Unit) or Oversight Organization Selection: Please select the CRU. OB/GYN The Clinical Research Unit that takes responsibility for this study. Please select Medicine as the CRU only if the PI is in one of these Divisions or Institutes: Endocrinology, Gastroenterology, General Internal Medicine, Geriatrics, Hematology, Infectious Diseases, Nephrology, Pulmonary, Rheumatology & Immunology, Center for Applied Genomics and Precision Medicine, Center for the Study of Aging and Human Development, Duke Molecular Physiology Institute. More information on CRUs can be found on the Duke Office of Clinical Research (DOCR) website, http://docr.som.duke.edu Questions concerning CRU selection should be directed to docr.help@dm.duke.edu. For questions about the Campus Oversight Organization, please visit Campus Oversight | |
| CRU (Clinical Research Unit) or Oversight Organization Selection: Please select the CRU. OB/GYN The Clinical Research Unit that takes responsibility for this study. Please select Medicine as the CRU only if the PI is in one of these Divisions or Institutes: Endocrinology, Gastroenterology, General Internal Medicine, Geriatrics, Hematology, Infectious Diseases, Nephrology, Pulmonary, Rheumatology & Immunology, Center for Applied Genomics and Precision Medicine, Center for the Study of Aging and Human Development, Duke Molecular Physiology Institute. More information on CRUs can be found on the Duke Office of Clinical Research (DOCR) website, http://docr.som.duke.edu Questions concerning CRU selection should be directed to docr.help@dm.duke.edu. For questions about the Campus Oversight Organization, please visit Campus Oversight | |

- If outside key personnel will have access to Duke PHI, a data transfer agreement AND external site IRB approval (or IRB authorization agreement) will be needed. See HRPP policy Use of Research Data by Former Duke Students or Former Duke Faculty and Employees
- In the panel below, "PHI" is Protected Health Information.

## Entry 1

| Name | Olola Oneko |
|---|---|
| Study Role | Study Physician |
| Email Address | ololaoneko@gmail.com |
| Institution / Organization | Kilimanjaro Christian Medical Centre (KCMC) |
| Will he/she have access to<br>Duke P.H.I.? | ○ Yes • No |
| Is he/she an unpaid<br>volunteer at Duke on the<br>study? | O Yes • No |

## **Indicate the Protocol source below:**

The protocol source is the author of the protocol. If the protocol is a joint authorship between multiple sources, select the primary author.

An IRB fee may be assessed for all research that is supported by for-profit entities and requires full board review. For additional information, see the **IRB fees section of the IRB web site** 

- PI initiated
- C Commercial / Industry (for-profit entity) initiated
- C Federal Government initiated
- Cooperative Group Initiated
- C Foundation (non-profit group) initiated
- Other

## **Sponsor and Funding Source**

## Add all funding sources for this study:

| Sponsor Name | Sponsor Type | Contract<br>Type: | Project<br>Number | Award<br>Number |
|---|---|---|---|---|
| Duke Endowment | Institutional | Grant | | |
| Name: | Duke Endowment | | | |
| Type: | Institutional | | | |
| Role: | Funding | | | |
| ontract Number: | | | | |
| Period: | From: to: | | | |
| ution the Primary Grant | No | | | |
| en who is the Primary<br>? | | | | |
| | Duke Endowment Name: Type: Role: ontract Number: Period: ution the Primary Grant en who is the Primary | Duke Endowment Name: Duke Endowment Type: Institutional Role: Funding ontract Number: Period: From: to: ution the Primary Grant No | Duke Endowment Institutional Name: Duke Endowment Type: Institutional Role: Funding Ontract Number: Period: Period: Type: No Sponsor Type Type: Type: Institutional Funding No Period: No No | Duke Endowment Institutional Name: Duke Endowment Type: Institutional Role: Funding Period: From: to: ution the Primary Grant Number Type: Number |

| Contract Type: | Grant | | | | |
|---|---|---|---|---|---|
| Project Number: | | | | | |
| Award Number: | | | | | |
| Grant Title: | Duke Global Health Fieldworl | < | | | |
| PI Name:<br>(If PI is not the same as identified<br>on the study.) | | | | | |
| Explain Any Significant Discrepancy: | | | | | |
| □ National Institutes of Health (NIH) | Externally Peer-Reviewed | Grant | 1R01CA195500-<br>01 | | |
| Sponsor Name: | National Institutes of Health | (NIH) | | | |
| Sponsor Type: | Externally Peer-Reviewed | | | | |
| Sponsor Role: | Funding | | | | |
| Grant/Contract Number: | 1R01CA195500-01 | | | | |
| Project Period: | From: to: | | | | |
| Is Institution the Primary Grant Holder: | Yes | | | | |
| Contract Type: | Grant | | | | |
| Project Number: | 1R01CA195500-01 | | | | |
| Award Number: | | | | | |
| Grant Title: | | | | | |
| PI Name:<br>(If PI is not the same as identified<br>on the study.) | | | | | |
| Explain Any Significant Discrepancy: | | | | | |
| Is this a federally funded study? | | | | | |
| ⊙ Yes O No | | | | | |
| Does this study have any of the fol | llowing? | | | | |
| <ul> <li>Industry sponsored protocol</li> <li>Industry funded Duke protocol</li> <li>Industry funded sub-contract f</li> <li>Industry provided drug/device</li> <li>SBIR/STTR funded protocol</li> </ul> | l<br>from another institution | | | | |
| C Yes • No | | | | | |
| As part of this study, will any samp<br>Sponsor, a Sponsor subcontractor, | | o/from Du | ike to/from anyo | ne other than | the |
| O Yes ⊙ No | | | | | |
| Is the Department of Defense (DO | D) a funding source? | | | | |

| O Yes ⊙ No | |
|---|---|
| For Federally funded studies: | |
| Is your funding subject to, and does it comply with, the funding agency's policy for data sharing? • Yes • No Check all that apply: | |
| <ul> <li>NIH Genome Sharing - dbGaP</li> <li>NIH Genome Sharing - GWAS</li> <li>NIH Genome Sharing - NCI databases</li> <li>NIH Genome Sharing - other</li> <li>Non-NIH Genomic</li> <li>✓ General Data Sharing</li> </ul> | |
| Enter the Grant Number or Other Federal Agency Proposal or Application Number: 1R01CA195500-01 | |
| Note: The Federal Funding Agency ID Number is the Sponsor's grant number assigned to your project and available on your Notice of Award (example: R01HL012345). | |
| If known, enter the SPS (Sponsored Projects System) number if applicable: | |
| <ul> <li>In the Initial Submission Packet, attach the following: <ol> <li>The entire grant, or an explanation of why a grant is not needed.</li> <li>NIH institutional Certificate form related to data sharing (if applicable).</li> </ol> </li> <li>The entire grant is needed so that it may be reviewed against the protocol for concordance.</li> </ul> | |
| Have you successfully synced your protocol to OnCore by clicking the 'Sync Data Over API' button at the of this page? | ne top |
| Please verify that the protocol has been created in OnCore before submitting this application for PI Signoff. | |
| <ul> <li>Yes, I synced my protocol to OnCore and verified it was successfully sent by logging into OnCore.</li> <li>I may have forgotten! I'll click it again right now, just to be sure, and verify it was successfully sent by logging into OnCore.</li> </ul> | |
| Mobile Devices and Software | |
| Does this study involve the use of a software or a mobile application? | |
| O Yes No | |
| List all software, including third party (non-Duke) and mobile apps, that will be utilized for ascertainm recruitment, or conduct of the research/project: (eg, MaestroCare, DEDUCE): | ent, |

| Multi-site Research |
|---|
| Is this a multi-site study? |
| Is the Duke PI/Co-PI the lead investigator or primary grant awardee? |
| ⊙ Yes O No |
| Is the primary grant awardee a Duke employee? |
| ⊙ Yes ○ No |
| Is a Duke employee the holder of the IND or IDE? |
| <ul><li>Yes</li><li>No</li><li>N/A</li></ul> |
| Is Duke the central coordinating center for this study? |
| ⊙ Yes O No |
| Is Duke serving as a central statistical center for this study? |
| O Yes ⊙ No |
| Is Duke serving as a central laboratory, reading center, analysis center or other central resource for this study? |
| ● Yes O No |
| Do you have ten or more sites? |
| O Yes ⊙ No |
| Complete for each site if Duke is the Primary grant awardee or coordinating center: |
| Entry 1 |
| Site Name: AIIMS |
| City: New Delhi |
| State/Province: |
| Country: India |

| | Site Contact Information |
|---|---|
| Primary Contact Name: | Neerja Bhatla |
| Primary Contact Phone: | |
| Primary Contact Email: | |
| , , , , , , , | neerja.bhatla07@gmail.com |
| | Site Details |
| Does the site have an IRB? | ⊙ Yes ○ No |
| Site IRB approval expiration | |
| date: | |
| If date not provided, explanation of why: | Approval letter given for the life of the study. No expiration. |
| Has the site granted | ⊙ Yes O No |
| permission for the research to be conducted? | |
| Does the site plan to rely on the DUHS IRB for review? | C Yes © No |
| What is the status of the | <b>⊙</b> Open |
| study at this site? | C Closed |
| Site approval letters or site | Attach site approval letters, site closure letterS (if applicable), or site |
| personnel lists: | personnel lists in the Initial Submission Packet. |
| Entry 2 | |
| Site Name: | Kenyatta University |
| City: | Nairobi |
| State/Province: | |
| Country: | Kanya |
| | Kenya |
| | Site Contact Information |
| Primary Contact Name: | Anthony Wanyoro |
| Primary Contact Phone: | |
| Primary Contact Email: | wanyara anthany@lay as l |
| | wanyoro.anthony@ku.ac.ke |
| | Site Details |
| Does the site have an IRB? | ⊙ Yes ○ No |
| | - 105 - NO |

| Site IRB approval expiration date: | 11/12/2016 |
|---|---|
| If date not provided, explanation of why: | |
| Has the site granted permission for the research to be conducted? | ⊙ Yes O No |
| Does the site plan to rely on the DUHS IRB for review? | O Yes ⊙ No |
| What is the status of the study at this site? | <ul><li>○ Open</li><li>⊙ Closed</li></ul> |
| Site approval letters or site personnel lists: | Attach site approval letters, site closure letterS (if applicable), or site personnel lists in the Initial Submission Packet. |

## Entry 3

| Site Name: | Kilimanjaro Christian Medical Centre |
|---|---|
| City: | Moshi |
| State/Province: | |
| Country: | Tanzania |
| | Site Contact Information |
| Primary Contact Name: | Bariki Mchome |
| Primary Contact Phone: | |
| Primary Contact Email: | barikimchome@gmail.com |
| | Site Details |
| Does the site have an IRB? | • Yes • No |
| Site IRB approval expiration date: | 03/25/2018 |
| If date not provided, explanation of why: | |
| Has the site granted permission for the research to be conducted? | ⊙ Yes ○ No |
| Does the site plan to rely on the DUHS IRB for review? | O Yes ⊙ No |
| What is the status of the study at this site? | Open Closed |
| Site approval letters or site personnel lists: | Attach site approval letters, site closure letterS (if applicable), or site personnel lists in the Initial Submission Packet. |

| | Site Contact Information |
|---|---|
| Country: | Zambia |
| State/Province: | Lusaka |
| City: | |
| Site Name: | University Teaching Hospital |
| Entry 5 | |
| personnel lists: | personnel lists in the Initial Submission Packet. |
| study at this site? Site approval letters or site | <ul> <li>○ Open</li> <li>ⓒ Closed</li> </ul> Attach site approval letters, site closure letterS (if applicable), or site |
| Does the site plan to rely on<br>the DUHS IRB for review?<br>What is the status of the | O Yes ⊙ No |
| Has the site granted permission for the research to be conducted? | • Yes O No |
| If date not provided, explanation of why: | |
| Site IRB approval expiration date: | 06/20/2017 |
| Does the site have an IRB? | ⊙ Yes ○ No |
| | Site Details |
| Filmary Contact Email: | ginovenegas@hotmail.com |
| Primary Contact Phone: Primary Contact Email: | |
| Primary Contact Name: | Gino Venegas |
| | Site Contact Information |
| Country: | Peru |
| State/Province: | |
| City: | Lima |
| Site Name: | Liga Peruana de lucha contra el cancer |

| | Groesbeck Parham |
|---|---|
| Primary Contact Phone: | |
| Primary Contact Email: | professorparham@gmail.com |
| | Site Details |
| Does the site have an IRB? | ⊙ Yes ○ No |
| Site IRB approval expiration date: | 04/07/2019 |
| If date not provided,<br>explanation of why: | |
| Has the site granted permission for the research to be conducted? | O Yes O No |
| Does the site plan to rely on the DUHS IRB for review? | O Yes ⊙ No |
| What is the status of the study at this site? | ○ Open Closed |
| Site approval letters or site personnel lists: | Attach site approval letters, site closure letterS (if applicable), or site personnel lists in the Initial Submission Packet. |
| Entry 6 | |
| Entry 6 Site Name: | Barranca clinic and San Rafael clinic |
| | Barranca clinic and San Rafael clinic |
| Site Name: | Barranca clinic and San Rafael clinic |
| Site Name: | |
| Site Name: City: State/Province: | |
| Site Name: City: State/Province: | Costa Rica |
| Site Name: City: State/Province: Country: | Costa Rica Site Contact Information |
| Site Name: City: State/Province: Country: Primary Contact Name: | Costa Rica Site Contact Information Alejandro Calderón |
| Site Name: City: State/Province: Country: Primary Contact Name: Primary Contact Phone: | Costa Rica Site Contact Information Alejandro Calderón n/a |

Site IRB approval expiration date:

If date not provided, explanation of why:

05/18/2021

| Has the site granted permission for the research to be conducted? | ⊙ Yes ○ No |
|---|---|
| Does the site plan to rely on the DUHS IRB for review? | |
| What is the status of the study at this site? | (•) ()nen |
| Site approval letters or site personnel lists: | ALLOCH SILE ODDIOVALIELLEIS, SILE CIOSULE IELLEIS HI ODDIICODIE I, OL SILE |
| | rocedures that will be used to inform sites of unanticipated problems in<br>terim results, protocol modifications and other information that may be<br>subjects: |
| Duke IRB procedures regarding the following will be adhered and reported to both Duke and external IRBs. Unanticipated problems will be reported to each site PI as soon as possible via telephone or email. Unanticipated problems will be promptly reported to both IRBs within ten business days of the investigator becoming aware of the event, study personnel will submit to the IRB a Notification of a Problem or Event Requiring Prompt Reporting to the IRB as A New Risk. The IRBs will be notified immediately (within 24 hours) upon learning of an unanticipated study-related death. | |
| How will you ensure that management, data analysis, and data safety and monitoring systems are adequate, given the nature of the research involved? | |
| The same procedures in the Duke IRB approved protocol will be followed. Members of the Duke University study team will perform the study at collaborating sites. They will ensure the same procedures are followed. | |
| How will you ensure that sample protocols and informed consent documents are developed and distributed to each collaborating institution? | |
| The study coordinator at Duke will develop and distribute the documents to all sites | |
| How will you ensure that each collaborating institution holds an applicable OHRP-approved Assurance? | |
| OHRP and FWA numbers can be verified here http://ohrp.cit.nih.gov/search/fwasearch.aspx? styp=bsc | |
| The FWA number for KCMC is FWA00002153 Kilimanjaro Christian Med College The FWA number for La Liga is FWA 15320 The FWA number for Nairobi is pending The FWA number for AIIMs is FWA00014191 | |

How will you ensure that each protocol is reviewed and approved by the IRB at the collaborating institution prior to the enrollment of subjects?

The study coordinator at Duke will verify this and make sure all approvals are uploaded to the Duke IRB prior to enrollment of subjects.

How will you ensure that any substantive modification by the collaborating institution of sample consent information related to risks or alternative procedures is appropriately justified?

The study coordinator at Duke and PIs will review all documents related to this study.

The FWA number for Zambia is FWA00000338

How will you ensure that informed consent is obtained from each subject in compliance with DHHS regulations?

A member of the Duke study team will be responsible for consenting patients and will be sure to be in compliance with DHHS regulations. Anyone obtaining informed consent will be required to take CITI training and Informed Consent Training. The local sites are responsible for compliance for those subjects enrolled.

## **Research Abstract**

## Please type your Research Abstract here:

The Research Abstract should summarize the main points of your study in one paragraph. The following guidelines may help you:

- 1. Purpose and objective (1-2 sentences)
- 2. Study activities and population group (2-4 sentences)
- 3. Data analysis and risk/safety issues (1-2 sentences)

Our goal is to bring the benefits of visual inspection with acetic acid with magnification (VIAM) to the primary screening setting in developing countries in an easy to use low-cost device, which we refer to as the transvaginal digital colposcope (TVDC). This device consists of a consumer grade digital camera found in the commonly used iPhone (Apple iPhone 4) and consumer grade light emitting diodes (LEDs) used in standard colposcopes, (Leisegang Optik 2), which all fit into the form factor of a tampon, a ubiquitous feminine hygiene product, and is significantly cheaper in cost to cervicography (standard of care used at two of the sites, Kilimanjaro Christian Medical Center (KCMC) and University Teaching Hospital (UTH)). The system comes with its own light source and requires significantly less training than cervicography as it can be simply be placed at the entrance to the speculum for image capture, without the need to adjust the light source or camera (focusing, positioning, etc). We will conduct pilot studies at multiple institutions where the goal will be to perform a side-by-side comparison of transvaginal colposcopy and the standard of care. In addition, to the clinical study objective, we will assess health provider acceptance, opinions, and experiences through pre- and post-transvaginal colposcopy surveys.

## **Research Summary**

## State your primary study objectives

Our goal is to bring the benefits of visual inspection with acetic acid with magnification (VIAM) to the primary screening setting in developing countries in an easy to use low-cost device, which we refer to as the transvaginal digital colposcope (TVDC). This device consists of a consumer grade digital camera found in the commonly used iPhone (Apple iPhone 4) and consumer grade light emitting diodes (LEDs) used in standard colposcopes, (Leisegang Optik 2), which all fit into the form factor of a tampon, a ubiquitous feminine hygiene product, and is significantly cheaper in cost to cervicography (standard of care used at these international sites. The system comes with its own light source and requires significantly less training than cervicography as it can be simply be placed at the entrance to the speculum for image capture, without the need to adjust the light source or camera (focusing, positioning, etc). We will conduct pilot studies at multiple institutions where the goal will be to perform a side-by-side comparison of transvaginal colposcopy and the standard of care. In addition, to the clinical study objective, we will assess health provider acceptance, opinions, and experiences through pre- and post-transvaginal colposcopy surveys.

## State your secondary study objectives

## Please select your research summary form:

Standard Research Summary Template

This is the regular (generic) research summary template which is required for all regular applications (unless your protocol fits under the other research summary templates in this category). Use of these instructions is helpful for ensuring that the research summary contains all necessary elements.

## **Standard Research Summary**

## **Purpose of the Study**

Objectives & hypotheses to be tested

We have developed a miniature colposcope called the transvaginal digital colposcope (TVDC). The system has been designed and constructed and will be used to obtain images of cervical tissue. The system is based on the same technology used in a traditional colposcope. This device consists of a consumer grade digital camera found in the commonly used iPhone (Apple iPhone 4 and other mobile phones) and consumer grade light emitting diodes (LEDs) used in standard colposcopes, (Leisegang Optik 2), which all fit into the form factor of a tampon, a ubiquitous feminine hygiene product, and is significantly cheaper in cost to cervicography (standard of care used at one of the study sites, The Kilimanjaro Christian Medical Center (KCMC)). The form factor of the device was inspired by an endotracheal intubation tube and digital tampon applicator. In this work, we will implement the TVDC ultimately intended for trans-vaginal use without the need for a speculum. **Figure 1** shows comparative images between a commercial clinical colposcope and our novel device collected from out Duke University protocol (pro00008173). **Figure 2** describes our novel transvaginal digital colposcope. The primary objective of this research is to establish concordance between our transvaginal digital colposcope and other standard of care screening techniques. Our secondary objective is physician assessment of the transvaginal digital colposcope.

**Fig. 1:** Digital image comparison with a Leisegang Optik 2 clinical digital colposcope (18 megapixel CMOS imager) at working distance of ~300mm and 7.5 magnification of 2 different cervixes under white light illumination (A) and green filter applied (B) versus the prototype transvaginal digital colposcope (2 MP CMOS imager) at working distance of between of 30-40 mm, for ~4X magnification, (Panel C and D), both with white LED illumination. Note, panels (A and C) and (B and D) are corresponding to the same cervix, with the clinical digital colposcope taking an image of the acetowhitened cervix followed by the transvaginal digital colposcope.

## **Background & Significance**

• Should support the scientific aims of the research

The most efficient strategy for prevention of cervical cancer in low and middle income countries is to screen using Human Papilloma Virus (HPV) testing or visual inspection with acetic acid (VIA), followed by treatment of pre-cancerous lesions using cryotherapy. In East Africa, where HPV testing is not routinely available, VIA or VIA with low power magnification (VIAM) is used to screen the population at a primary health care level, and VIA/VIAM combined with cryotherapy or LEEP is performed at some primary and secondary and all tertiary health centers. Significant concerns about embarrassment and pain due to screening from the speculum, gender of the health provider, privacy and distance to the screening center are some of the main reasons why women do not get screened. Another important issue with VIA/VIAM is its low specificity compared to the Pap smear. We believe that the operational scaling (labor costs) and issues with acceptability of screening to be major impediments to creating widespread cervical cancer prevention in Tanzania and other developing countries. Our program strives to address these issues by delivering a high-volume, cost-effective cervical cancer screening solution for low resource environments, through partnerships with the following institutions:

- 1. Duke University Medical Center, Durham, NC
- 2. Kilimanjaro Christian Medical Center (KCMC) in Moshi, Tanzania. Closed as of 2021
- 3. Cancer Institute WIA, Chennia, India
- 4. Liga Peruana de lucha contra el cancer, Lima, Peru Closed as of 2021
- 5. Kiambu Hospital, Kenya
- 6. All India Institute of Medical Sciences (AIIMS), New Delhi, India
- 7. University Teaching Hospital Lusaka, Zambia Closed as of 2021
- 8. Barranca clinic and San Rafael clinic within the Seguro Social network

We have IRB approval with Liga Peruana de lucha contra el cancer in Lima, Peru and with Kilimanjaro Christian Medical Centre (KCMC). We have therefore included those approvals and consent forms. The other sites will be added through amendments as the studies are approved. Based on our current IRB approvals, the total enrollment is 500 subjects (200 at Liga Peruana, 100 at KCMC, 100 at AIIMS, 50 at UTH).

With the addition of Costa Rica, we will be increasing the enrollment by 800. Target enrollment should be completed over an 18-month period. Therefore the new enrollment as of December 2020 will be 1400. Of note, our collaboration with Costa Rica is via IARC not a specific clinic within the country. We will not be consenting subjects for our study. We will be receiving de-identified images only. We are in the process of working on a DTA with their site. No enrollment as of 4-19-2021.

## **Design & Procedures**

• Describe the study, providing detail regarding the study intervention (drug, device, physical procedures, manipulation of the subject or the subject's environment, etc.). Discuss justifications for placebo control, discontinuation or delay of standard therapies, and washout periods if applicable. Identify procedures, tests and interventions performed exclusively for research purposes or more frequently than standard of care. Include alternative therapies, concurrent therapies discontinued per protocol, risk benefit ratio, and use of tissue/specimens. Discuss monitoring during washout periods if applicable. Include brief description of follow-up, if any.

**Fig.3:** Gaumard Zoe Gynecologic Simulator used for in-vitro prototype development and for field training health providers.

In this multi-site clinical study, we will compare images collected with our TVDC to the standard of care at each collaborating institution. Patients undergoing cervical cancer screening or LEEP for the treatment of premalignant cervical dysplasia will be enrolled into the study. We will recruit 50-100 patients at each site, including DUMC. Before implementation of the clinical protocol, all health providers will be trained on the use of the transvaginal colposcope using a life-sized mannequin (Gaumard Zoe Gynecologic Simulator

S504.100) with different cervices (healthy, dysplastic) (**Fig. 3**). This will include implementation of the colposcope and operation of the laptop or tablet to acquire images and positioning of the colposcope to optimize image quality. In addition, training in sterilization of device in between patients, maintenance, and daily quality control will be conducted.

The clinical protocol will be as follows. Each enrolled patient will undergo the standard of care for cervical cancer screening at each institution followed by the TVDC. The standard of care for each institution is provided below.

ISAI n t c msaea tint g t di e uacs ti r A a odcc noiq f d ui cur ase r e d e d fr ао s m s st t a a n n d d a a r r d d o o f f c са a r r e e ? ?

UCYY ni o e e v l s sер rs o it s у с Мо ер di y С al С е n t е

r

```
Ki C Y Y
li e e e
mrss
a v
nj ic
ао
r g
o r
Са
h p
ri h
st y
ia
n
Μ
е
di
С
al
С
е
n
t
е
r
\mathsf{C} \mathsf{V} \mathsf{Y} \mathsf{N}
a is e o
n us (c
са
      а
e l
      m
r I
       er
I n
       а
n s
       n
st p
       ot
it e
      u
ис
      S
t ti
      е
е о
       d
Wn
       )
I w
A it
  h
  Α
  С
  е
  ti
  С
  Α
  ci
  d
Li C Y Y
goee
alss
Рр
е о
r s
ис
ао
n p
ау
d
е
lu
С
h
а
```

С О n tr а el С а n С е r Ki V Y N a is e o m u s b a u l ΗΙ o n s s рі р t e al c ti 0 n W it h Α С е ti С Α ci d AVYNII is e o Mus S a Ţ Ι n S р е С ti 0 n W it h а С е ti С а ci d U C ni e

rs ic e e it o S S y g Т r e a a p c h hi y n g Н 0 S рi t al

After screening with standard of care, then images will be acquired with the TVDC. Research procedures will be carried out with the use of the speculum. Speculum-free implementation will be addressed in a future study. Twenty to forty images will be captured with the TVDC at a rate of 5-15 frames per second. Twenty to forty images will be captured in order to allow for the auto focus mechanism to capture a focused image with the transvaginal colposcope. At maximum, this will add 2 minutes to the patient procedure. Imaging with the TVDC may be repeated during the same visit for until satisfactory (focused, full view of cervix) images are acquired. If biopsies are necessary, as per standard of care, they will be collected from suspicious sites. Research biopsies will not be collected nor will this study cover biopsy costs. Biopsy must be done after imaging because bleeding at the site of biopsy may interfere with the digital images.

All physicians and healthcare workers who perform screening for this study will be asked to complete the following:

- 1. The clinical evaluation table for both the standard of care and transvaginal colposcope. This will be completed once for each patient. This table is included under the full protocol section.
- 2. A survey before beginning the clinical work with the transvaginal colposcope. This will be completed once for each healthcare worker. This survey is included under the full protocol section.
- 3. A survey after study completion to assess acceptance, opinions, and experiences with the system. This will be completed once for each healthcare worker. The pre- and post- assessment surveys are included in the Appendix. This survey is included under the full protocol section.
- 4. A mobile phone survey
- 5. In addition, members of the healthcare team and hospital staff will be asked think aloud questions and mobile landscape questions.

## **Selection of Subjects**

• List inclusion/exclusion criteria and how subjects will be identified.

The population will include those who are undergoing cervical cancer screening for the diagnosis of cervical cancer. Specific criteria are below:

#### Inclusion criteria

Patients undergoing cervicography OR colposcopy OR VIA OR patients undergoing LEEP for the treatment of cervical cancer.

- Age 25 and greater
- Patients of all ethnic will be included.
- Ability to understand and the willingness to sign a written informed consent document.

#### **Exclusion Criteria**

• Children and subjects under 25.

Since the study poses no discernible risk to a pregnant woman or an unborn fetus, therefore pregnant patients will be included in this research. Our transvaginal colposcope is currently being used in another DUMC research study where pregnant women are eligible to participate. That research study is pro00008173.

## **Subject Recruitment and Compensation**

• Describe recruitment procedures, including who will introduce the study to potential subjects. Describe how you will ensure that subject selection is equitable and all relevant demographic groups have access to study participation (per 45 CFR 46.111(a) (3)). Include information about approximately how many DUHS subjects will be recruited. If subjects are to be compensated, provide specific prorated amounts to be provided for expenses such as travel and/or lost wages, and/or for inducement to participate.

One of the local collaborating doctors will identify subjects who are eligible for the study from their patient population. The physician (or nurse) will introduce the study to potential subjects and, if they agree to be contacted, the nurse or a research team member will explain the purpose and background of the study, the selection criteria, the patient's involvement, benefits, risks, compensation (for injury), costs, alternatives, confidentiality and disclosure issues with the patient. All external sites may not have research coordinators to perform this step; therefore may be performed by a nurse. Informed written consent will be obtained from patients who are willing to participate at the time of the screening or LEEP visit. Information from each patient's medical record will be recording, including but not limited to cervical pathology, age and menopausal status. Table 1 shows a sample table of patient demographical information to be collected. HIV status will be recorded because cervical dysplasia is known to progress faster in HIV positive women and it is therefore important to record. A total 200 patients will be recruited for the study. HIV status is critical information to collect in this study because the progression from low grade to high grade to cancer is faster with patients that are HIV positive. We anticipate the ideal screening method for cervical cancer screening would be HPV status, HIV status and screening with the TVDC. A sample size of 50-100 patients at each site should allow for the potential examination of at least 10 patients who have a positive screening (based on the occurrence of positive women in the cervical cancer screening programs). Each participating site will retain their original signed informed consent documents. Duke University will not obtain copies of informed consent from the collaborating institutions.

#### **Consent Process**

• Complete the consent section in the iRIS Submission Form.

## **Subject's Capacity to Give Legally Effective Consent**

• If subjects who do not have the capacity to give legally effective consent are included, describe how diminished capacity will be assessed. Will a periodic reassessment occur? If so, when? Will the subject be consented if the decisional capacity improves?

Subjects who are not competent to give consent will not be included.

## **Study Interventions**

• If not already presented in #4 above, describe study-related treatment or use of an investigational drug or biologic (with dosages), or device, or use of another form of intervention (i.e., either physical procedures or manipulation of the subject or the subject's environment) for research purposes.

The patient's procedure will be carried out according to standard of care. In addition, the trans-vaginal colposcope will be used to collect digital images of the cervix.

## **Risk/Benefit Assessment**

• Include a thorough description of how risks and discomforts will be minimized (per 45 CFR 46.111(a) (1 and 2)). Consider physical, psychological, legal, economic and social risks as applicable. If vulnerable populations are to be included (such as children, pregnant women, prisoners or cognitively impaired adults), what special precautions will be used to minimize risks to these subjects? Also identify what available alternatives the person has if he/she chooses not to participate in the study. Describe the possible benefits to the subject. What is the importance of the knowledge expected to result from the research?

The risk of placing the trans-vaginal colposcope in the vagina is no greater than the risk of performing a Pap smear. The system's outer shell is made out of medical grade ABS plastic with a biocompatible heat shrink tubing sleeve made of PTFE or similar material for enhanced waterproofing and protection. Medical grade and biocompatible adhesives (Loctite 4011) are used to seal the device and prevent infiltration of water and bodily fluids. Excess body fluids are first removed with a Super Sani-Cloth Germicidal wipe and then the following the standard sterilization procedure (immersion in 2% hydrogen peroxide solution or 10% bleach solution). A fresh Supersani Germicidal wipes are wrapped around probes to keep them sterile between patients. The edges of the probe face are also chamfered to avoid a sharp edge so there should be minimal risk of puncture caused by the probe with the pressure exerted. The device does not emit ultraviolet light and emits only visible light from 400 to 700 nm and has been tested to pose minimal eye and tissue risk per IESNA RP-27 and ANSI/IEC 60825-1 LED safety standards. The device is electrically isolated from the body. Heating of the tissue due to light exposure is minimal and can be neglected compared to much less in magnitude from the heat generated by conventional halogen illumination sources used in traditional clinical colposcopes due to the utilization of more efficient LEDs. Optical information obtained through the images will not affect decisions regarding the treatment of the patient because it will be analyzed at a later time. Participants may experience mild discomfort during use of the probe and there may be risks unknown at this time.

## **Costs to the Subject**

• Describe and justify any costs that the subject will incur as a result of participation; ordinarily, subjects should not be expected to pay for research without receiving direct benefit.

There are no costs to subjects as a result of participating in this research.

## **Data Analysis & Statistical Considerations**

Describe endpoints and power calculations. Provide a detailed description of how study data will be
analyzed, including statistical methods used, and how ineligible subjects will be handled and which
subjects will be included for analysis. Include planned sample size justification. Provide estimated time
to target accrual and accrual rate. Describe interim analysis including plans to stop accrual during
monitoring. Phase I studies, include dose escalation schema and criteria for dose escalation with
definition of MTD and DLT.

Lesions observed with the transvaginal colposcope and the standard of care will be assessed using the clinical evaluation table of endpoints included in the full protocol section of the IRB submission. In addition, we will compare image quality from the data in the clinical evaluation table that compared transvaginal colposcopy and standard of care screening. Note that visual inspection with acetic acid (VIA) does not require the use of a camera we will therefore be unable to compare images collected to the TVDC to the standard of care for sites using only VIA. For the sites that use VIA only, we will compare the responses from the clinical evaluation table which includes questions such as: 1) can you see aceto-whitening, 2) can you see vasculature, 3) can you see a lesion. For a full list of questions, see the clinical evaluation table in Section 7, Full Protocol.

Statistical comparisons between TVDC and standard of care (SOC) images will be done using paired t-tests (pairs of TVDC and SOC outcomes on the same patient), with non-parametric adjustments, based on clinical evaluation table and other outcomes such as procedure time as dependent variables (with N=48 to 50 patients). For example, we postulate that the difference between mean scores (TVDC-SOC) will be positive, against the null hypothesis that they are the same. We expect approximately 3-4 physicians to implement SOC and TVDC on the same patients with about 12 to 16 patients available per physicians. We will also compare TVDC and SOC using a repeated-measure ANOVA (implemented using a linear mixed effect model) to account for physician effect. Due to low number of physicians available for our study, we will treat physician effect as a fixed effect. Alternatively, a simple regression one-way ANOVA model can also be fitted by using the difference scores between TVDC and SOC as the dependent variable where physicians are entered as a 3 or 4-level categorical/group variable (between-patients effect). An overall significance level of 0.050 will be used for statistical tests (type III Wald t-tests).

**Physician variability:** Our primary outcome measure will be the quadratic weighted Kappa [4, 5] statistic for concordance. Furthermore, cluster adjusted by site and/or clinician) analysis can be used to address nested stepwise logistic regression model will be used to determine potential factors for disconcordant interpretation of the cervical images using both a backward and forward entry model using a  $p_r$  value of 0.15 backward selection and  $p_e$  value of 0.10 for forward selection, respectively in the STATA statistical software package.

Should we suspect excessive between-physician variability, we will conduct sensitivity analyses by treating physicians as random-effects (with pairs of outcomes on the same patient nested within physicians) under a range of intra-class correlation coefficients postulated to account for between-physician heterogeneity (equivalent to varying physician random-effect variance over a suitable range). Note that, ignoring physician variability, a sample size of 50 achieves 80% power to detect a Cohen's d of 0.41 (a moderate effect size) with a significance level (alpha) of 0.050 using a two-sided Wilcoxon test assuming that the actual distribution is normal.

## **Data & Safety Monitoring**

• Summarize safety concerns, and describe the methods to monitor research subjects and their data to ensure their safety, including who will monitor the data, and the frequency of such monitoring. If a data monitoring committee will be used, describe its operation, including stopping rules and frequency of review, and if it is independent of the sponsor (per 45 CFR 46.111(a) (6)).

A Data & Safety Monitoring team will not be used, however, the DUMC Institutional Review Board (IRB) will be responsible for monitoring the clinical study for its compliance to National Commission for the Protection of Human Subjects of Biomedical and Behavioral Research entitled: *Ethical Principles and Guidelines for the Protection of Human Subjects of Research*. The researchers will be responsible for reporting any Adverse Events (AEs) and any protocol deviations to the IRB by submitting the appropriate paperwork to the IRB. The protocol will also be reviewed and approved by each site's Institutional Review Board.

| Similar protocols for this research have already been submitted, reviewed and approved by DUMC'S IRB. The protocols are reviewed on an annual basis and amendments to the protocol may be written at any time should there be new personnel associated with the research, major/minor changes to the research proposal (including changes in PHI and consent forms) or any other change to the protocol that must be made to reflect the actual research that is being performed. | |
|---|---|
| Duke is the Coordinating Center for this multi-site study. Duke and the study team are committed to the protection of all subjects enrolled into this study. The study coordinator, Marlee Krieger, will be responsible for promptly reporting important study information to all sites. The PIs of each site will be included on the correspondence including any and all coordinators. This will be done electronically via email with send receipt confirmation. Important information includes unanticipated problems involving risks to subjects or others, interim results and protocol modifications. In addition, the email updates, regular meetings will be held via teleconference. This will be done on approximately a monthly basis. Finally, site visits will also be made to each location on average annually. | |
| Privacy, Data Storage & Confidentiality | |
| Complete the Privacy and Confidentiality section of the iRIS submission form. | |
| Describe Role of External Personnel: | |
| n/a | |
| Study Scope | |
| Does this study have a cancer focus? Cancer focus includes studies that enroll >50% oncology or mathematology patients; or, preventing, detecting, and diagnosing cancer or understanding the impact of cancer on patients and their caretakers. | _ |
| Does this study have a cancer focus? Cancer focus includes studies that enroll >50% oncology or ma hematology patients; or, preventing, detecting, and diagnosing cancer or understanding the impact of | _ |
| Does this study have a cancer focus? Cancer focus includes studies that enroll >50% oncology or mathematology patients; or, preventing, detecting, and diagnosing cancer or understanding the impact of cancer on patients and their caretakers. | _ |
| Does this study have a cancer focus? Cancer focus includes studies that enroll >50% oncology or mathematology patients; or, preventing, detecting, and diagnosing cancer or understanding the impact of cancer on patients and their caretakers. O Yes O No | _ |
| Does this study have a cancer focus? Cancer focus includes studies that enroll >50% oncology or mathematology patients; or, preventing, detecting, and diagnosing cancer or understanding the impact of cancer on patients and their caretakers. O Yes O No Are you using a drug, biologic, food, or dietary supplement in this study? | f |
| Does this study have a cancer focus? Cancer focus includes studies that enroll >50% oncology or mathematology patients; or, preventing, detecting, and diagnosing cancer or understanding the impact of cancer on patients and their caretakers. O Yes No Are you using a drug, biologic, food, or dietary supplement in this study? O Yes No Are you using a medical device, an algorithm (whether computer based or not), an in vitro diagnostic | f |
| Does this study have a cancer focus? Cancer focus includes studies that enroll >50% oncology or mathematology patients; or, preventing, detecting, and diagnosing cancer or understanding the impact of cancer on patients and their caretakers. ○ Yes No Are you using a drug, biologic, food, or dietary supplement in this study? ○ Yes No Are you using a medical device, an algorithm (whether computer based or not), an in vitro diagnostic using samples to look for biomarkers in this study? | f |
| Does this study have a cancer focus? Cancer focus includes studies that enroll >50% oncology or manatology patients; or, preventing, detecting, and diagnosing cancer or understanding the impact of cancer on patients and their caretakers. ○ Yes No Are you using a drug, biologic, food, or dietary supplement in this study? ○ Yes No Are you using a medical device, an algorithm (whether computer based or not), an in vitro diagnostic using samples to look for biomarkers in this study? ○ Yes No | f |
| Does this study have a cancer focus? Cancer focus includes studies that enroll >50% oncology or manatematology patients; or, preventing, detecting, and diagnosing cancer or understanding the impact of cancer on patients and their caretakers. ○ Yes No Are you using a drug, biologic, food, or dietary supplement in this study? ○ Yes No Are you using a medical device, an algorithm (whether computer based or not), an in vitro diagnostic using samples to look for biomarkers in this study? ○ Yes No Does this study involve a Humanitarian Use Device (HUD)? | test, or |

| Does this study specify or require the performance of diagnostic procedures using ionizing radiation ( DEXA, CT scans, nuclear medicine scans, etc.) that are beyond the standard of care? | x-rays, |
|---|---|
| O Yes ⊙ No | |
| Does this study specify or require the performance of therapeutic procedures using ionizing radiation (accelerator, brachytherapy or systemic radionuclide therapy) that are beyond the standard of care? | |
| O Yes No | |
| Will the participant be subjected to increased or decreased ambient pressure? | |
| O Yes ⊙ No | |
| Do you plan to recruit subjects from Duke Regional Hospital (DRH)? | |
| O Yes ⊙ No | |
| Do you plan to recruit subjects from Duke Raleigh Hospital (DRAH)? | |
| O Yes No | |
| Does this study utilize the Duke Early Phase Clinical Research Unit (DEPCRU)? | |
| ○ Yes • No | |
| Are you using the Duke logo in any advertisements? | |
| Are you using the Duke logo in any advertisements? O Yes • No | |
| O Yes | |
| O Yes | |
| <ul> <li>○ Yes</li></ul> | oduct |
| Is this study retrospective, prospective, or both? "Retrospective" means that data or samples already in existence (collected prior to the study submission) will be used. "Prospective" means there will be data or samples collected in this study for research purposes. Retrospective Prospective Prospective Retrospective and Prospective Retrospective and Prospective Retrospective and Prospective New retrospective and prospective: Is this a review soley of information collected for non-research purposes (i.e. a review of medical records)? Yes No Does this protocol include any research using botulinum toxin, including the FDA-approved clinical process. | oduct |
| Is this study retrospective, prospective, or both? "Retrospective" means that data or samples already in existence (collected prior to the study submission) will be used. "Prospective" means there will be data or samples collected in this study for research purposes. Retrospective Prospective Retrospective Retrospective and Prospective If the study is both retrospective and prospective: Is this a review soley of information collected for non-research purposes (i.e. a review of medical records)? Yes ○ No Does this protocol include any research using botulinum toxin, including the FDA-approved clinical pro(Botox)? | oduct |

| <ul> <li>Any cells that have been modified by a viral vector</li> <li>Any other genetically-modified cells</li> <li>Any genetically-modified virus, bacterium, or other agent</li> <li>Any other recombinant or synthetic nucleic acid</li> </ul> |
|---|
| O Yes • No |
| Subject Population Groups and Enrollment |
| Population Groups (Select <u>targeted</u> population groups only): |
| Note: |
| <ul> <li>If Minors are included, the study will be routed to the Department of Pediatrics for Pediatric Risk Assessment.</li> <li>Students and Employees over whom Key Personnel have a supervisory role may not be enrolled in this study</li> </ul> |
| ✓ Adults Minors who are Wards of State Minors Duke Patients Pregnant Women Fetuses Prisoners Adults incapable of giving consent Adults with diminished capacity Handicapped subjects Students Employees Healthy Controls Deceased subjects Blanket Protocol |
| Please select any population groups excluded from participation in this study: |
| ☐ Pregnant women |
| Maximum number of subjects to be consented at Duke: |
| Enter a single number. If you anticipate consenting a range of subjects, enter the <b>upper</b> limit of the range. The number should represent the maximum number of subjects for the life of the study. 50 |
| Maximum number of subjects to be consented at all sites: |
| Enter a single number. If you anticipate consenting a range of subjects, enter the <b>upper</b> limit of the range. The number should represent the maximum number of subjects for the life of the study. 1400 |
| Subject Procedures and Costs |
| Biobank - Does this study involve the collection, use, tracking, banking (storage) or distribution of human biological specimens? |

| Check all the apply: Genetic Testing Genetic Testing Genetic Reportable Infectious Diseases Human Cell Banking Use of Human Embryonic Stem Cells Use of Human-induced Pluripotent Stem Cells Use of Other Cells Derived from Human Embryos Use of Human-Induced Pluripotent Stem Cells Use of Both Fluids Use of Other Cells Derived from Human Embryos Use of Other Cells Derived from Human Embryos Use of Human Tissue Use of Blood (or its components) Not Applicable Will blood be drawn in this study for research purposes? Yes O No Will the Operating Room be used in this study? Include only research time, not clinical care time. Yes No Will there be extra costs to subjects or insurance as a result of the research (e.g. tests, hospitalization)? Yes No Will there be Subject Compensation? Yes No Subject Recruitment Materials For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. All materials that will be used to advertise the study in order to recruit subjects must be approved by the IRB. | Human biological specimens include blood or its components, healthy or diseased tissue, bodily fluids, DNA /RNA or human stem cells. | |
|---|---|---|
| Check all the apply: Genetic Testing Genet Transfer DNA Banking Testing for Reportable Infectious Diseases Human Cell Banking "Use of Human-Induced Pluripotent Stem Cells "Use of Human-Induced Pluripotent Stem Cells "Use of Human-Induced Pluripotent Stem Cells "Specialized Cell Populations for Cell Therapy Use of Human Tissue Use of Bodily Fluids Use of Bodily Fluids Use of Bodily Fluids Will blood be drawn in this study for research purposes? Yes ② No Will the Operating Room be used in this study? Include only research time, not clinical care time. Yes ② No Will there be extra costs to subjects or insurance as a result of the research (e.g. tests, hospitalization)? Yes ③ No Will there be Subject Compensation? Subject Recruitment Materials For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | O Yes ⊙ No | |
| Genetic Testing Gene Transfer DNA Banking Testing for Reportable Infectious Diseases Human Cell Banking *Use of Human Embryonic Stem Cells *Use of Human-Induced Pluripotent Stem Cells *Use of Other Cells Derived from Human Embryos *Use of Other Cells Derived from Human Embryos *Use of Bodily Fluids Use of Bodily Fluids Use of Bodily Fluids Use of Bodily Fluids Use of Bodily Fluids Use of Bodily Fluids Will blood be drawn in this study for research purposes? Yes ® No Will the Operating Room be used in this study? Include only research time, not clinical care time. Yes ® No Will there be extra costs to subjects or insurance as a result of the research (e.g. tests, hospitalization)? Yes ® No Will there be Subject Compensation? Yes ® No Subject Recruitment Materials For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | Procedures | |
| Genetic Testing Gene Transfer DNA Banking Testing for Reportable Infectious Diseases Human Cell Banking *Use of Human Embryonic Stem Cells *Use of Human-Induced Pluripotent Stem Cells *Use of Other Cells Derived from Human Embryos *Use of Other Cells Derived from Human Embryos *Use of Bodily Fluids Use of Bodily Fluids Use of Bodily Fluids Use of Bodily Fluids Use of Bodily Fluids Use of Bodily Fluids Will blood be drawn in this study for research purposes? Yes ® No Will the Operating Room be used in this study? Include only research time, not clinical care time. Yes ® No Will there be extra costs to subjects or insurance as a result of the research (e.g. tests, hospitalization)? Yes ® No Will there be Subject Compensation? Yes ® No Subject Recruitment Materials For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | Check all the apply: | |
| Gene Transfer DNA Banking Testing for Reportable Infectious Diseases Human Cell Banking "Use of Human Embryonic Stem Cells "Use of Human Induced Pluripotent Stem Cells "Use of Human/Animal Chimeric Cells "Sepecialized Cell Populations for Cell Therapy Use of Human Insue Use of Bodily Fluids Use of Bilood (or its components) Not Applicable Will blood be drawn in this study for research purposes? Yes | | |
| DNA Banking Testing for Reportable Infectious Diseases Human Cell Banking *Use of Human Embryonic Stem Cells *Use of Human Induced Pluripotent Stem Cells *Use of Human Induced Pluripotent Stem Cells *Use of Human Induced Pluripotent Stem Cells *Use of Human Insue Use of Bodily Fluids Use of Bodily Fluids Use of Bodily Fluids Use of Bodily Fluids Will blood be drawn in this study for research purposes? Yes No Will the Operating Room be used in this study? Include only research time, not clinical care time. Yes No Will there be extra costs to subjects or insurance as a result of the research (e.g. tests, hospitalization)? Yes No Will there be Subject Compensation? Yes No Subject Recruitment Materials For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | | |
| Testing for Reportable Infectious Diseases Human Cell Banking "Use of Human Embryonic Stem Cells "Use of Human Embryonic Stem Cells "Use of Other Cells Derived from Human Embryos "Use of Other Cells Derived from Human Embryos "Use of Human-Infimation Cell Therapy Use of Bodily Fluids Use of Bodily Fluids Use of Bodily Fluids Use of Bodily Fluids Use of Blood (or its components) Will blood be drawn in this study for research purposes? C Yes | | |
| Human Cell Banking "Use of Human Embryonic Stem Cells "Use of Human Embryonic Stem Cells "Use of Other Cells Derived from Human Embryos "Use of Other Cells Derived from Human Embryos "Use of Human/Animal Chimeric Cells "Specialized Cell Populations for Cell Therapy Use of Bodily Fluids Use of Blood (or its components) Not Applicable Will blood be drawn in this study for research purposes? Yes | | |
| *Use of Human Embryonic Stem Cells *Use of Human-Induced Puripotent Stem Cells *Use of Human-Induced Puripotent Stem Cells *Use of Human/Animal Chimeric Cells *Specialized Cell Populations for Cell Therapy Use of Blood (or its components) Will be of Blood (or its components) Not Applicable Will blood be drawn in this study for research purposes? Yes | | |
| *Use of Human-induced Pluripotent Stem Cells *Use of Other Cells Derived from Human Embryos *Use of Other Cells Derived From Human Embryos *Use of Human/Ainnal Chimeric Cells *Specialized Cell Populations for Cell Therapy Use of Bollod (or its components) Vestor of Blood (or its components) Not Applicable Will blood be drawn in this study for research purposes? Yes | | |
| *Use of Other Cells Derived from Human Embryos *Use of Human/Animal Chimeric Cells *Specialized Cell Populations for Cell Therapy Use of Blood (or its components) Will blood be drawn in this study for research purposes? Will blood be drawn in this study for research purposes? Will the Operating Room be used in this study? Include only research time, not clinical care time. Yes No Will there be extra costs to subjects or insurance as a result of the research (e.g. tests, hospitalization)? Yes No Will there be Subject Compensation? Yes No Subject Recruitment Materials For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | | |
| *Use of Human/Animal Chimeric Cells *Specialized Cell Populations for Cell Therapy Use of Human Tissue Use of Bodily Fluids Use of Bodily Fluids Use of Blood (or its components) Not Applicable Will blood be drawn in this study for research purposes? Yes | | |
| *Specialized Cell Populations for Cell Therapy Use of Human Tissue Use of Bood (or its components) Not Applicable Will blood be drawn in this study for research purposes? Yes No No | | |
| Use of Blood (or its components) Use of Blood (or its components) Not Applicable Will blood be drawn in this study for research purposes? C Yes | | |
| Use of Bodily Fluids Use of Blood (or its components) Not Applicable Will blood be drawn in this study for research purposes? Yes No Will the Operating Room be used in this study? Include only research time, not clinical care time. Yes No Will there be extra costs to subjects or insurance as a result of the research (e.g. tests, hospitalization)? Yes No Will there be Subject Compensation? Yes No Subject Recruitment Materials For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | | |
| Use of Blood (or its components) Not Applicable Will blood be drawn in this study for research purposes? Yes No Will the Operating Room be used in this study? Include only research time, not clinical care time. Yes No Will there be extra costs to subjects or insurance as a result of the research (e.g. tests, hospitalization)? Yes No Will there be Subject Compensation? Yes No Subject Recruitment Materials For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | Use of Bodily Fluids | |
| Will the Operating Room be used in this study? Include only research time, not clinical care time. Yes No Will there be extra costs to subjects or insurance as a result of the research (e.g. tests, hospitalization)? Yes No Will there be Subject Compensation? Yes No Subject Recruitment Materials For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | Use of Blood (or its components) | |
| Will the Operating Room be used in this study? Include only research time, not clinical care time. ○ Yes No Will there be extra costs to subjects or insurance as a result of the research (e.g. tests, hospitalization)? ○ Yes No Will there be Subject Compensation? ○ Yes No Subject Recruitment Materials For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | ✓ Not Applicable | |
| Will the Operating Room be used in this study? Include only research time, not clinical care time. ○ Yes No Will there be extra costs to subjects or insurance as a result of the research (e.g. tests, hospitalization)? ○ Yes No Will there be Subject Compensation? ○ Yes No Subject Recruitment Materials For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | Will blood be drawn in this study for research purposes? | |
| Include only research time, not clinical care time. Ores No Will there be extra costs to subjects or insurance as a result of the research (e.g. tests, hospitalization)? Ores No Will there be Subject Compensation? Ores No Subject Recruitment Materials For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | O Yes © No | |
| Will there be extra costs to subjects or insurance as a result of the research (e.g. tests, hospitalization)? ○ Yes No Will there be Subject Compensation? ○ Yes No Subject Recruitment Materials For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | Will the Operating Room be used in this study? | |
| Will there be extra costs to subjects or insurance as a result of the research (e.g. tests, hospitalization)? ○ Yes No Will there be Subject Compensation? ○ Yes No Subject Recruitment Materials For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | Include only research time, not clinical care time | |
| Will there be extra costs to subjects or insurance as a result of the research (e.g. tests, hospitalization)? ○ Yes No No No No No No No No | | |
| Will there be Subject Compensation? ○ Yes No Subject Recruitment Materials For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | O Yes • No | |
| Will there be Subject Compensation? ○ Yes No Subject Recruitment Materials For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | Will there be extra costs to subjects or insurance as a result of the research (e.g. tests, hospitalization | n)? |
| Subject Recruitment Materials For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | O Yes ⊙ No | |
| Subject Recruitment Materials For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | | |
| Subject Recruitment Materials For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | Will there be Subject Compensation? | |
| For each document to be reviewed, use the table below to provide the following information: Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | C Yes ⓒ No | |
| Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | Subject Recruitment Materials | |
| Attach a copy of each advertisement that you will be using with this study in the Initial Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | | |
| Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | For each document to be reviewed, use the table below to provide the following information: | |
| | Submission Packet. If any Ad will have multiple wording variations, attach a copy of each version of the Ad. | |

| Types of subject recruitment materials include, but are not limited to, the following: | | | | |
|---|---|---|---|---|
| Direct Advertising Posters Billboards Flyers Brochures | | | | |
| Media Advertising Newspaper Ads Magazine Ads Radio Ads TV commericals / Video Internet website Social Media | | | | |
| Other Types of Advertise Newsletter Email Postcards / Letters | | | | |
| (Note: Doctor-to-Doctor le | etters do not require 1RB a | approvar) | | |
| Document name | Material category | Location material displayed | Has this material previously been approved by the IRB? | |
| No records have been a | dded | • | | |
| | | Consent Process | | |
| Attach draft consent fo | orms in the Initial Revi | ew Submission Packet. | | |
| Consent forms must be M download a copy of the co | | ollow the specific format outli | ined by the IRB. <u>Click here</u> to | |
| | . Those fields will be used | | Continuing Review form when it is approved by the | |
| Who will conduct the c | onsent process with p | rospective participants? | | |
| Give the person's role in this study (PI, Study Coordinator, etc.): | | | | |
| The study coordinator or | Duke study team membe | er will obtain informed cons | sent. | |
| Who will provide conse | ent or permission? | | | |
| (Select all that apply): | | | | |
| Participant | | | | |
| ☐ Parent(s) or Legal Guardian(s) ☐ Legally Authorized Representative (LAR) | | | | |
| Legally Authorized Re | presentative (LAK) | | | |
| How much time will th approached about part | | nt (or legally authorized | representative) have between b | peing |

| If you are not giving the person overnight to consider whether or not to participate, please justify. The study coordinator or Duke study team member will obtain informed consent. | |
|---|---|
| Where will the consent process occur? | |
| Patients will not be consented in public. The consent process will occur in a private room with the patient. | |
| What steps will be taken in that location to protect the privacy of the prospective participant? | |
| Patients will not be consented in public. Consent will be obtained in a private room with a door that shuts. | |
| How much time will be allocated for conducting the initial consent discussion, including presenting the information in the consent document and answering questions, with each prospective participant? | |
| Due to the diagnostic nature of this study, patients must be consented day of the procedure. Patients will be given about an hour to decide whether or not to participate. | |
| What arrangements will be in place for answering participant questions before and after the consent is signed? | |
| The study will first be introduced to the patient by a member of their healthcare team. If they agree to be contacted, a clinic nurse (not a member of the research team), or a member of the study team will explain the purpose, background of the study, the selection criteria, the patient's involvement, benefits, risks, compensation, costs, alternatives, confidentiality, and disclosure issues with the patient. If a patient is interested then written consent will be obtained from them at the time of screening or LEEP visit. The study team and specifically those obtaining consent are prepared to answer any study related questions. Participants are encouraged to ask questions at any time. A study team member OR the physician is available to answer questions before or after the consent is signed. | |
| Describe the steps taken to minimize the possibility of coercion or undue influence. | |
| Since patients must consent the day of their procedure, the study team will attempt to make sure that each potential participant has as much time as needed to considered participating in the study. It is also made clear that there is no benefit or rewards for participation. Compensation will not be offered. | |
| What provisions will be in place to obtain consent from participants who do not read, are blind or who do no read/understand English? | t |
| The consent form will be translated in the primary language of each country with a participating institution. | |
| Do you plan to obtain written consent for the conduct of research? | |
| ⊙ Yes O No | |
| Protected Health Information (PHI) | |
| Indicate how you intend to use potential subjects' Protected Health Information (PHI): | |
| <ul> <li>I will review, but not record, PHI prior to consent.</li> <li>I will record PHI prior to consent.</li> <li>I do not intend to use PHI prior to consent.</li> <li>I will record PHI without consent. (decedent research, database repository, chart review)</li> </ul> | |

| Describe the specific PHI that will be reviewed to prepare a research protocol and/or to ascertain and/or recruit subjects: | | | | | |
|---|---|---|---|---|---|
| Various eligibility criteria will be verified prior to consent included age and procedure | | | | | |
| Principal Investigator's Affirmation: | | | | | |
| The PHI is | he PHI is necessary for the purposes of this activity. | | | | |
| ⊙ Yes C | Yes O No | | | | |
| The PHI w | ne PHI will be used solely for this activity. | | | | |
| ⊙ Yes C | No | | | | |
| The PHI w | ill not leave DUHS. | | | | |
| ⊙ Yes C | ) No | | | | |
| The PHI w | ill not be written down or re | corded | prior to the subject si | gning a research cons | ent form. |
| ⊙ Yes C | No | | | | |
| | se the information accessed on or publication. | throug | gh this RPR procedure | for any other purpose | , including for |
| ⊙ Yes C | No | | | | |
| | | | Devices | | |
| Include a | II devices being evaluate | d in th | nis study: | | |
| information<br>any Human | devices being evaluated in to<br>a about a humanitarian use on<br>itarian Use Device that does<br>product labeling and its safet | device<br>s not re | where requested.Also equire an IDE because | dd devices without an | IDE here, including |
| Complete a<br>Packet. | an <u>IDE Billing Notice</u> as appli | icable. | This can be attached | with the Brochure in th | ne Initial Submission |
| | | | | Will the device to be evaluated or | IDE |
| View<br>Details | Device Name | | Is the Device FDA<br>Approved | the Humanitarian Use Device be manufactured at Duke? | /Compassionate<br>Use Request<br>Number |
| | ☐ Transvaginal digital colposcope | | No | Yes | Abbreviated |
| Device S | Device Source Duke | | е | | |
| CMS Category | | . □ B | | | |
| | Is the device provided to subject free of charge? | | | | |
| | his a HUD (HDE)? | | | | |
| HDE Number | | | | | |
| Is the Device FDA Approved | | No | | | |
| Will the device to be evaluated or | | | | | |

the Humanitarian Use Device be

manufactured at Duke?

Yes

| Do you have an IDE number for this device? | Yes |
|---|---|
| IDE/Compassionate Use Request<br>Number | Abbreviated |
| IDE Holder | PI holds the IDE |
| IDE Details | The FDA determined this to be an abbreviated IDE so there is no IDE number Due to programming issues, the correct response is "NO" to the question, "Will the device to be evaluated or the Humanitarian Use Device be manufactured at Duke?" |
| In the opinion of the sponsor, select the level of risk associated with this device | No Significant Risk |

Who will be responsible for the storage, inventory and control of the device to be evaluated or the Humanitarian Use Device?

Dr. Nimmi Ramanujam

Where will the device to be evaluated or the Humanitarian Use Device be stored?

Dr. Nimmi Ramanujam's lab

Who will be responsible for giving or administering the device to be evaluated or the Humanitarian Use Device to the research subject?

The PI or key personnel

From where will the device to be evaluated or the Humanitarian Use Device be dispensed?

Gross Hall

At the completion of this research study, what will be done with the unused or returned device or the Humanitarian Use Device?

The device will be returned to Duke.

## **Privacy and Confidentiality**

## Explain how you will ensure that the subject's privacy will be protected:

Consider privacy interests regarding time and place where subjects provide information, the nature of the information they provide, and the type of experience they will be asked to participate in during the research.

We are committed to maintaining patient confidentiality. Patient data will always be entered using a patient identification number. To protect against the risk of loss of confidentiality, the study will follow the procedures specified by the DUMC Institutional Review Board and Institutional Review Boards of the other centers for maintaining confidentiality. Data will be stored in a locked, secure location.

## Describe how research data will be stored and secured to ensure confidentiality:

How will the research records and data be protected against inappropriate use or disclosure, or malicious or accidental loss or destruction? Records and data include, for example, informed consent documents, case

report forms or study flow sheets, survey instruments, database or spreadsheets, screening logs or telephone eligibility sheets, web based information gathering tools, audio/video/photo recordings of subjects, labeled specimens, data about subjects, and subject identifiers such as social security number.

Data will be stored in a locked, secure location. Computerized data is accessible only by password, and a centralized monitoring system records and reports all access to data. CRFs will be identified by study number only to insure subject anonymity. The link between the unique subject number and the subject's identity will be maintained in a secure location at the research site. No subject identifiers will be used in the presentation of data. Study records that identify subjects will be kept confidential as required by law. Subjects will be informed that their study physician and his/her study team will report the results of study related tests to the PI and to the sponsor. Subjects will be informed that their records may be reviewed in order to meet federal or state regulations. Reviewers may include the FDA, IRBs, or the NIH. Subjects will be informed that if their research record is reviewed, their entire medical record may also need to be reviewed.

## **Application Questions Complete**

## Please click Save & Continue to proceed to the Initial Submission Packet.

The Initial Submission Packet is a short form filled out after the protocol application has been completed. This is an area to attach protocol-related documents, consent forms, and review the application.